CLINICAL TRIAL: NCT01951547
Title: The Effect of Non-surgical Periodontal Therapy on Host Response and Microbiological Profile of Type 2 Diabetics With Periodontal Disease.
Brief Title: The Periodontal Disease and Diabetes Mellitus Interrelationship Among Adult Malaysians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Rathna Devi Vaithilingam, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMRG344/11HTM
Record Dates: First submitted 2013-08-30; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes
Keywords: HbA1c; hs-CRP; non-surgical periodontal therapy; oral health education; probing pocket depth; plaque index; gingival bleeding index.
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nonsurgical periodontal therapy (Experimental): Nonsurgical periodontal therapy given at baseline
  Interventions: Procedure: Nonsurgical periodontal therapy; Procedure: Oral hygiene instructions
- Oral hygiene instructions (Active Comparator): Oral hygiene instructions given at baseline
  Interventions: Procedure: Oral hygiene instructions

INTERVENTIONS:
Procedure: Nonsurgical periodontal therapy — Periodontal intervention All patients were instructed in oral hygiene methods using a soft bristled toothbrush, a compact-tuft toothbrush, interdental brushes and dental floss utilizing the modified Bass technique. Full mouth debridement, which consisted of scaling and root planing, was done in a single visit for all subjects using an ultrasonic scaler and gracey curettes. Additionally, all patients were given a 0.12% Chlorhexidine mouthrinse (Hexipro®). They were instructed to rinse three times a day using 15ml each time for a period of 14 days commencing immediately after completion of full mouth debridement. Thereafter at each recall visit, all participants were re-motivated and professional prophylaxis was performed.
  Arms: Nonsurgical periodontal therapy
Procedure: Oral hygiene instructions — All patients were instructed in oral hygiene methods using a soft bristled toothbrush, a compact-tuft toothbrush, interdental brushes and dental floss utilizing the modified Bass technique.

SUMMARY:
Periodontitis, a chronic inflammatory disease which results in irreversible attachment loss, bone destruction and tooth loss, is a major oral health problem affecting 90.2% of Malaysian population. It was initially demonstrated that Type 2 Diabetes (T2D) was a risk factor for periodontitis and subsequently a two-way relationship between diabetes and periodontitis was proposed. Diabetes has been shown to cause defects in neutrophil function by overproduction of pro-inflammatory mediators such as Tumour necrosis factor-α, Interleukin-1β and Prostaglandin E2 by macrophages. The inflammatory mediators released in response to plaque have been reported to be insulin antagonists that disturb binding of insulin to its receptors and further complicate hyperglycaemia in T2D. The hyperglycaemia in diabetics promotes more pathogenic bacteria into the subgingival microenvironment making them more susceptible to chronic periodontitis. Studies however differ in the types of periodontal pathogens present in these pockets. At the same time, very few studies have quantified them. This study proposes to investigate the effect that non-surgical periodontal therapy (NSPT) has on the periodontal parameters, HbA1c levels, microbiological profile and CRP levels of T2D patients with chronic periodontitis as compared to oral hygiene education (OHE)alone.

DETAILED DESCRIPTION:
Ethical approval was obtained from both the Medical Ethics Boards of University Malaya Medical Centre (MEC Ref No: 696.9) and University Malaya Dental Centre [DF PE1002/0045(P)]. One hundred and twelve type 2 diabetic patients (diagnosed at least 1 year prior to the study) between ages of 30 to 70 were screened from the outpatient Diabetes Clinic of the University Malaya Medical Centre and a total of 40 patients who fulfilled the inclusion and exclusion criteria were recruited for the study. The recruited patients were then registered at the Periodontology Clinic at the Faculty of Dentistry, University of Malaya. Patient information sheets regarding the study and verbal explanations were given to all patients. Informed consent was obtained from all recruited patients with the understanding that they could withdraw from the study at any time. Screening and treatment of patients commenced from January 2010 till December 2011.

The sample size calculation determined that 15 subjects per treatment arm would provide 80% power to detect a minimum difference of 1% (11.0 mmol/mol) change in HbA1c between test and control. Accordingly, a sample of 20 subjects per arm (40 in total) was recruited to compensate for possible drop-outs during the study period.

All patients were randomly assigned via a coin toss to age matched NSPT and OHE groups. Investigator 1 screened and enrolled participants and assigned them to age-matched groups. Investigator 2 performed the random allocation sequence using coin toss method to assign participants to the different interventions while Investigator 1 performed all intervention. There was no blinding of participants or examiner.

As only one examiner was involved in the study, intra-examiner reliability assessment was executed to validate the ability of the examiner to constantly reproduce the quantitative outcome measurements of the clinical parameters used. The Plaque Index (PI), Gingival Bleeding Index (GBI), Probing Pocket Depth (PPD) and Probing Attachment Loss (PAL) were measured in the time interval of about 3 hours. Utilizing Kappa statistics, good agreements (>0.8) were obtained for reproducibility of all recorded clinical parameters.

All recruited patients underwent full periodontal assessment at baseline, 2 months after assigned treatment and 3 months after assigned treatment. The clinical examination included Plaque Index (PI), Gingival Bleeding Index (GBI), Probing Pocket Depth (PPD) and Probing Attachment Loss (PAL) measured with an electronic constant- force probe (Florida Probe®).

All patients were instructed in oral hygiene methods using a soft bristled toothbrush, a compact-tuft toothbrush, inter-dental brushes and dental floss utilizing the modified Bass technique. Full mouth debridement, which consisted of scaling and root planing, was done in a single visit for all subjects in the NSPT group using an ultrasonic scaler and Gracey curettes. Additionally, all patients in the NSPT group were given a 0.12% Chlorhexidine mouthrinse (Hexipro®). They were instructed to rinse three times a day using 15ml each time for a period of 14 days commencing immediately after completion of full mouth debridement. Thereafter at each recall visit, all participants were re-motivated and professional prophylaxis was performed on those in the test group.

15 ml of venous blood was collected from each patient at baseline, prior to treatment and at 3 months after assigned treatments. Levels of glycosylated haemoglobin (HbA1c) and systemic hs-C-Reactive Protein (hs-CRP) were assessed. Hs-CRP levels were assessed using tests for high sensitivity CRP (hs-CRP). All blood investigations were done at a private laboratory (Gnosis Laboratories Sdn. Bhd) with no affiliation to the Department of Periodontology. The HbA1c testing is DCCT aligned and the Quality Assurance of the laboratory is certified under Bio-Rad Laboratories (USA), EQAS (External Quality Assurance Services).

Deepest pockets were identified (minimum 5 pockets with PPD ≥ 5 mm) and isolated with cotton rolls. This was followed by careful removal of supragingival plaque using cotton pellets and curettes. Subgingival plaque samples were subsequently collected using sterile curettes and pooled into sterile DNAse-free and RNase-free polyethylene tube containing 1ml Phosphate Buffer Solution (PBS) and frozen at -800C until commencement of q-PCR analysis.

Automated DNA extraction was performed in the lab using the QIAcube machine (Qiagen®). 100 µl of plaque sample was placed in a 1.5 ml centrifuge tube and was centrifuged at a speed of 5,000 × g for 10 minutes on a tabletop centrifuge machine to obtain a pellet. The pellets were then placed on the QIAcube-shaker for automated DNA extraction by QIAcube machine using DNeasy® Blood & Tissue Mini Kit and QIAmp® DNA accessory set. All reagents provided in the kit were manually placed into the reagent bottle rack in the machine prior to the start of the process. Finally, the "Bacterial DNA" protocol was selected from the machine's protocol list. Briefly, the Qiacube machine underwent five consecutive steps which included lysis, incubate, bind, wash and elution processes. At the end of the process, 100µl of eluted DNA was available. The extracted DNA were then tested for concentration and purity using Nanodrop machine. The DNA was then stored in -80⁰C before bacterial identification using q-PCR machine.

The concentration and purity of extracted DNA was determined using the spectrophotometer machine (Thermo Scientific NanoDrop™ 2000 Spectrophotometers) which was connected with a PC based software. 0.1 µl of eluted DNA was pipetted onto the lower pedestal arm. A fiber optic cable (the receiving fiber) is embedded within this pedestal. A second fiber optic cable (the source fiber) located in the upper pedestal arm is then brought into contact with the liquid sample causing the liquid to bridge the gap between the ends of the two fibers. A pulsed xenon flash lamp provides the light source and a spectrometer utilizing a linear CCD array analyzes the light passing through the sample. The DNA concentration from both plaque samples and reference strain were measured and recorded accordingly. The extracted DNAs were eventually stored in -20⁰C until the commencement of q-PCR procedure.

The detection and quantification of P. gingivalis, A.actinomycetemcomitans, P.intermedia and T.forsythia from plaque samples were done using Applied Biosystems® 7500 Real-Time PCR Systems which was connected to PC based software. The quantification was done by projecting the cycle threshold (Ct) value of the samples on the standard curve of the known amount (concentration) of bacteria reference strain.

For this purpose, a known amount of extracted DNA of the bacteria was serially diluted (10 fold dilution) and was subjected to RT-PCR amplification. This was done to provide a standard curve prior to amplification of DNA from plaque samples using q-PCR. Optimization was carried out in order to get the optimum standard curve for quantification. A final 10 fold dilution standard curve of reference strains (range from 10ng/µl- 0.0001 ng/µl) with R2 value of 0.956 was used as a base for quantification.

To determine the sensitivity of the q-PCR technique, serial samples containing known concentrations of individual microorganisms were processed for q-PCR analysis. The lowest concentration that resulted in a positive PCR product was regarded as the sensitivity of the assay.

q-PCR amplification was done in a total reaction mixture volume of 20µl. This mixture contained 2µl of purified DNA from plaque sample/ reference strain to act as PCR template, 10 µl of 2x TaqMan® Fast Advanced Master Mix (PCR buffer, dNTP's, Amplitaq Gold, reference signal, uracil N-glycosylase, MgCl2; Applied Bio systems, Foster City, CA, USA), 1µl Custom Taqman® Gene Expression Assay (20x) and 7µl nuclease-free water. The procedures were conducted using 96-well reaction plates.

All the components of the reaction mixture (except DNA sample) were added onto a 1.5mL micro centrifuge tube. The tube was capped and vortexed briefly. The tubes were then centrifuged to spin down the contents and eliminate air bubbles. The mixture was then transferred to a 96 well reaction plate and followed by addition of 2µl DNA sample. The reaction plate was then covered with optical adhesive cover after the entire well had been occupied. This reaction plate was again briefly centrifuged to spin down the content and to ensure all bubbles were eliminated.

This mixture was then subjected to an initial amplification cycle of 50ºC for 2 minutes and 95ºC for 10 minutes, followed by 45 cycles at 95ºC for 15s and 60ºC for 1 minute. The q-PCR amplification plot for each sample was analyzed to determine the Ct value. The Ct value was then projected to the standard curve of reference strain for the quantification.

Comparisons of changes in PI, GBI, PPD(%) and PAL (%) both within and between the groups were performed using the chi-square test. Intragroup comparison for mean PPD, mean PAL, mean HbA1c, mean CRP and frequency of detection of P. gingivalis, A.actinomycetemcomitans, P.intermedia and T.forsythia were assessed with the paired sample t-test whereas intergroup comparisons for the same variables was accomplished using an independent sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients whose diagnosis had been established (World Health Organization, 1999) and were on regular follow-ups for a minimum of 6 months.
* Patients should have at least 12 teeth present
* Patients with 2 or more interproximal sites (not on same tooth) with probing pocket depths of 5mm or more and 2 or more interproximal sites (not on same tooth)of probing attachment loss of 4mm or more which bled on probing.

Exclusion Criteria:

* Patients who had history of systemic antibiotic usage over the previous 4 months
* Patients who were pregnant
* Patients who had received non-surgical periodontal treatment within the past 6 months
* Patients who had received surgical periodontal treatment within the past 12 months
* Patients who were smokers
* Patients with a history of stroke or an acute cardiovascular event over the previous 12 months.
* Patients who had their diabetic medication changed during the course of the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effect of periodontal intervention on plaque score levels in diabetics with periodontal disease | Changes from baseline to 3 months
  Plaque score levels were evaluated at baseline, 2- and 3-months intervals
Effect of periodontal intervention on gingival bleeding index of diabetics with periodontal disease | Changes from baseline to 3 months
  Gingival bleeding index levels were evaluated at baseline, 2- and 3-months intervals
Effect of periodontal intervention on probing pocket depths of diabetics with periodontal disease | Changes from baseline to 3 months
  Probing pocket depths were evaluated at baseline, 2- and 3-months intervals
Effect of periodontal intervention on probing attachment levels of diabetics with periodontal disease | Changes from baseline to 3 months
  Probing attachment levels were evaluated at baseline, 2- and 3-months intervals

SECONDARY OUTCOMES:
Effect Of periodontal intervention on microbiological profile of diabetics with periodontal disease | Changes from baseline to 3 months
  Quantitative polymerase chain reaction (q-PCR) was used to determine the presence and levels of P. gingivalis, A. actinomycetemcomitans, P. intermedia and T. forsythia at baseline and 3 months follow up.
Effect of periodontal intervention on HbA1c levels of diabetics with periodontal disease | Changes from baseline to 3 months
  HbA1c levels were evaluated at baseline, 2- and 3-months intervals
Effect Of periodontal intervention on hs-CRP levels in diabetics with periodontal disease | Changes from baseline to 3 months
  HbA1c levels were evaluated at baseline and 3-months intervals

CONTACTS AND LOCATIONS:
Overall Officials: Rathna D Vaithilingam, MClinDent, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Taiyeb-Ali TB, Raman RP, Vaithilingam RD. Relationship between periodontal disease and diabetes mellitus: an Asian perspective. Periodontol 2000. 2011 Jun;56(1):258-68. doi: 10.1111/j.1600-0757.2010.00370.x. No abstract available. PMID 21501247
- [Background] Taylor GW, Borgnakke WS. Periodontal disease: associations with diabetes, glycemic control and complications. Oral Dis. 2008 Apr;14(3):191-203. doi: 10.1111/j.1601-0825.2008.01442.x. PMID 18336370
- [Background] Taylor GW, Burt BA, Becker MP, Genco RJ, Shlossman M, Knowler WC, Pettitt DJ. Severe periodontitis and risk for poor glycemic control in patients with non-insulin-dependent diabetes mellitus. J Periodontol. 1996 Oct;67(10 Suppl):1085-93. doi: 10.1902/jop.1996.67.10s.1085. PMID 8910827
- [Background] Boutaga K, van Winkelhoff AJ, Vandenbroucke-Grauls CM, Savelkoul PH. Comparison of real-time PCR and culture for detection of Porphyromonas gingivalis in subgingival plaque samples. J Clin Microbiol. 2003 Nov;41(11):4950-4. doi: 10.1128/JCM.41.11.4950-4954.2003. PMID 14605122
- [Background] Boutaga K, van Winkelhoff AJ, Vandenbroucke-Grauls CM, Savelkoul PH. The additional value of real-time PCR in the quantitative detection of periodontal pathogens. J Clin Periodontol. 2006 Jun;33(6):427-33. doi: 10.1111/j.1600-051X.2006.00925.x. PMID 16677332
- [Derived] Raman RP, Taiyeb-Ali TB, Chan SP, Chinna K, Vaithilingam RD. Effect of nonsurgical periodontal therapy verses oral hygiene instructions on type 2 diabetes subjects with chronic periodontitis: a randomised clinical trial. BMC Oral Health. 2014 Jun 25;14:79. doi: 10.1186/1472-6831-14-79. PMID 24965218